CLINICAL TRIAL: NCT00000969
Title: A Prospective, Randomized, Open-Label, Comparative Trial of Dideoxyinosine (ddI) Versus Dideoxycytidine (ddC) in HIV-Infected Patients Who Are Intolerant of or Who Have Failed Zidovudine (AZT) Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: CPCRA 002; 11554 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Didanosine; Drug Evaluation; Zidovudine
MeSH Terms: conditions — HIV Infections | interventions — Zalcitabine; Didanosine

INTERVENTIONS:
Drug: Zalcitabine
Drug: Didanosine

SUMMARY:
To evaluate and compare the effectiveness and toxicity associated with didanosine ( ddI ) and zalcitabine ( dideoxycytidine; ddC ) in patients with HIV infection who are intolerant of or have failed zidovudine ( AZT ) therapy.

Alternative and less toxic treatments need to be investigated for the treatment of HIV infection. Studies have shown that the dideoxynucleosides ddI and ddC may be effective antiretroviral agents in the treatment of HIV-infected individuals. However, ddI and ddC have yet to be compared on the basis of patient survival, drug tolerance, immunologic and virologic effectiveness, and the incidence of opportunistic infection or opportunistic malignancy. Results of this study will yield information regarding the relative therapeutic benefits and toxicities of each drug while providing alternative treatment to patients who are unable to tolerate or have had progression of disease while on AZT.

DETAILED DESCRIPTION:
Alternative and less toxic treatments need to be investigated for the treatment of HIV infection. Studies have shown that the dideoxynucleosides ddI and ddC may be effective antiretroviral agents in the treatment of HIV-infected individuals. However, ddI and ddC have yet to be compared on the basis of patient survival, drug tolerance, immunologic and virologic effectiveness, and the incidence of opportunistic infection or opportunistic malignancy. Results of this study will yield information regarding the relative therapeutic benefits and toxicities of each drug while providing alternative treatment to patients who are unable to tolerate or have had progression of disease while on AZT.

After baseline screening, patients are randomized to one of two treatment arms (ddI or ddC). Subjects are evaluated biweekly for the first 4 weeks of study, at 2 months, and every other month thereafter. Three dose levels of ddI (based on patient's weight at study entry) are compared with two dose levels of ddC (also based on patient weight). Patients who reach a new progression-of-disease primary endpoint after at least 12 weeks of treatment or a drug intolerance endpoint have the option of switching over to the alternate study drug; however, participants are encouraged to remain on their original drug assignment whenever possible. For any switchover, patients must be off the originally assigned drug for at least 72 hours before switching. Only one switchover is allowed.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Acyclovir (if patient is also receiving ddC, clinical monitoring should be more frequent).
* Analgesics, antiemetics, antidiarrheal agents, or other necessary treatment for symptomatic therapy.
* Interferons for maintenance therapy of Kaposi's sarcoma.
* GM-CSF.

Required:

* Prophylaxis against Pneumocystis carinii pneumonia (PCP) if their absolute CD4+ lymphocyte count is < 200 cells/mm3 at study entry. PCP prophylaxis for patient with CD4+ counts between 200 and 300 cells/mm3 is at discretion of patient's primary physician.
* NOTE: There is potential interaction of ddI and dapsone.

Concurrent Treatment:

Allowed:

* Transfusion, erythropoietin.

Patients must have the following:

* Zidovudine (AZT) failure after having received a cumulative duration of at least 6 months.
* AZT intolerance - rechallenge is not required for patients exhibiting = or > grade III cutaneous symptoms.
* Diagnosis of AIDS or CD4+ = or < 300 cells/mm3 OR AIDS-defining illness other than Kaposi's sarcoma.
* Willingness and ability to comply with protocol.
* Informed consent must be obtained for all study participants in accordance with state law, local IRB requirements, and 45 CFR Part 46. AMENDED 11/19/90 to include assent by minors if they are physically able, in addition to consent by parents.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Any disorders for which the study drugs are contraindicated (didanosine (ddI)) is contraindicated in renal impairment, heart disease, receiving renal dialysis.
* Active opportunistic infection.

Concurrent Medication:

Excluded:

* Other antiretroviral agents.
* Use of drugs associated with peripheral neuropathy or use of agents that may cause pancreatitis including intravenous pentamidine and alcohol should be restricted or avoided.

Concurrent Treatment:

Excluded:

* Other concurrent antiretroviral clinical trials.

Patients with the following are excluded:

* History of pancreatitis, peripheral neuropathy, uncontrolled seizures, renal impairment, heart disease, stage 2 or higher ADC.
* Any other disorders for which the study drugs are contraindicated, i.e., ddI is contraindicated in renal impairment, patients receiving renal dialysis, and heart disease.
* Receiving acute therapy for active AIDS defining opportunistic infection on enrollment.

Prior Medication:

Excluded:

* Didanosine (ddI).
* Dideoxycytidine (ddC) .

Excessive alcohol use that, in investigator's opinion, puts patient at risk of developing pancreatic disease.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Study Completion 1992-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kaplan C, Study Chair; Crane L, Study Chair; Abrams D, Study Chair
Locations (16):
- United States (16):
  - Community Consortium of San Francisco, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Hill Health Corp, New Haven, Connecticut
  - Wilmington Hosp / Med Ctr of Delaware, Wilmington, Delaware
  - Veterans Administration Med Ctr / Regional AIDS Program, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Comprehensive AIDS Alliance of Detroit, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Clinical Directors Network of Region II, New York, New York
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Richmond AIDS Consortium, Richmond, Virginia

REFERENCES:
- [Background] Bjorling LE, Hodges JS. Rule-based ranking schemes for antiretroviral trials. Stat Med. 1997 May 30;16(10):1175-91. doi: 10.1002/(sici)1097-0258(19970530)16:103.0.co;2-g. PMID 9179982
- [Background] Hogan CH, Hodges JS, Mugglin A, Peterson PM, Abrams DI, Saravolatz L. The perils of visit-driven endpoints in antiretroviral trials. Int Conf AIDS. 1996 Jul 7-12;11(1):237 (abstract no TuB522)
- [Background] Fleming TR, Neaton JD, Goldman A, DeMets DL, Launer C, Korvick J, Abrams D. Insights from monitoring the CPCRA didanosine/zalcitabine trial. Terry Beirn Community Programs for Clinical Research on AIDS. J Acquir Immune Defic Syndr Hum Retrovirol. 1995;10 Suppl 2:S9-18. PMID 7552519
- [Background] Goldman AI, Carlin BP, Crane LR, Launer C, Korvick JA, Deyton L, Abrams DI. Response of CD4 lymphocytes and clinical consequences of treatment using ddI or ddC in patients with advanced HIV infection. J Acquir Immune Defic Syndr Hum Retrovirol. 1996 Feb 1;11(2):161-9. doi: 10.1097/00042560-199602010-00007. PMID 8556398
- [Background] Abrams D, Goldman A, Launer C, Korvick J, Crane L, Deyton L. Results of a randomized open-label comparison trial of ddI and ddC in HIV infected patients who are intolerant of or have failed ZDV therapy; CPCRA 002. The Terry Beirn Community Programs for Clinical Research on AIDS. Int Conf AIDS. 1993 Jun 6-11;9(1):67 (abstract no WS-B24-4)
- [Background] Abrams DI, Goldman AI, Launer C, Korvick JA, Neaton JD, Crane LR, Grodesky M, Wakefield S, Muth K, Kornegay S, et al. A comparative trial of didanosine or zalcitabine after treatment with zidovudine in patients with human immunodeficiency virus infection. The Terry Beirn Community Programs for Clinical Research on AIDS. N Engl J Med. 1994 Mar 10;330(10):657-62. doi: 10.1056/NEJM199403103301001. PMID 7906384
- [Derived] Soeiro-de-Souza MG, Bio DS, David DP, Rodrigues dos Santos D Jr, Kerr DS, Gattaz WF, Machado-Vieira R, Moreno RA. COMT Met (158) modulates facial emotion recognition in bipolar I disorder mood episodes. J Affect Disord. 2012 Feb;136(3):370-6. doi: 10.1016/j.jad.2011.11.021. Epub 2012 Jan 4. PMID 22222175